CLINICAL TRIAL: NCT03761940
Title: An Observational Study Assessing the Health Status in Women With Early Breast Cancer, Treated With Breast Conserving Surgery and Radiotherapy
Brief Title: Health Status of Women With Breast Cancer
Acronym: OSTaRa
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 18/0059
Record Dates: First submitted 2018-10-26; First posted 2018-12-03 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Women With Early Breast Cancer; Breast Conserving Surgery; Radiotherapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Disease free: Women who have been treated for early breast cancer with breast conserving surgery and radiotherapy and at the time of completing study questionnaires are disease free.
  Interventions: Other: EQ5D questionnaire and a demographic questionnaire
- Local recurrences: Women who have been treated for early breast cancer with breast conserving surgery and radiotherapy and at the time of completing study questionnaires have been diagnosed with local recurrence and may be undergoing treatment for this.
  Interventions: Other: EQ5D questionnaire and a demographic questionnaire
- Distant disease: Women who have been treated for early breast cancer with breast conserving surgery and radiotherapy and at the time of completing study questionnaires have been diagnosed with distant disease and may be undergoing treatment for this.
  Interventions: Other: EQ5D questionnaire and a demographic questionnaire
- Mastectomy: Women who have been treated for early breast cancer with breast conserving surgery and radiotherapy and at the time of completing study questionnaires have undergone a mastectomy.
  Interventions: Other: EQ5D questionnaire and a demographic questionnaire

INTERVENTIONS:
Other: EQ5D questionnaire and a demographic questionnaire — questionnaires

SUMMARY:
The quality-adjusted life-year (QALY) is the outcome measure of choice in England and Wales for National Institute for Health and Care Excellence (NICE). To be able to conduct a cost utility analysis, QALY data is required. This can either be collected within trial or published data can be used.

In the United Kingdom (UK) there is no up to date QALY data for women with early breast cancer treated with surgery followed by radiotherapy. The OSTaRa Study aims to provide up to date QALY data for women in this cohort.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Over 18 year of age
* Has had breast cancer, treated with both breast conserving surgery and radiotherapy.
* Is willing to complete an EQ5D and a demographic questionnaire.

Exclusion Criteria:

* Does not speak sufficiently to complete a study questionnaires.
* Has not already been approached to complete an OSTaRa questionnaire.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Participants who satisfy the inclusion exclusion criteria can be selected either from clinic notes, MDT records, or at clinic.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-03-14 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
Questionnaire | 12 months
  Each subject will complete an EQ5D questionnaire, to allow Quality of Life to be calculated. The EQ5D uses a Likert scale which assesses five states (mobility, self care, usual care, pain and discomfort and anxiety and depression) at five different levels - none, slight, moderate, severe or unable to perform. Levels are coded 1-5 and a total score is then generated. Results for the demographic measured will be displayed as a percentage value.

CONTACTS AND LOCATIONS:
Locations (1):
- Great Western Hospitals NHS Foundation Trust, Swindon, Wiltshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The OSTaRa study team will adhere to SITU's data sharing policy.
Supporting Information: Study Protocol, ICF
Time Frame: Once the study has been published
Access Criteria: Apply to SITU requesting the study data set. Send your request to situ.trial@ucl.ac.uk
URL: http://www.ucl.ac.uk/situ